CLINICAL TRIAL: NCT01738425
Title: A Double-Blind, Placebo Controlled, Phase I Study to Assess Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Oral Doses of GIC-1001 in Normal Healthy Volunteers
Brief Title: A Clinical Phase I Study on GIC-1001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: gicare Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIC P2-458
Record Dates: First submitted 2012-11-23; First posted 2012-11-30 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Colonic Diseases
Keywords: GIC-1001; opioid agonist; sulfide; colonoscopy; gicare; Phase I; safety; tolerability; pharmacokinetics; healthy subjects; single ascending dose; multiple ascending dose; SAD; MAD; food effect
MeSH Terms: conditions — Colonic Diseases | interventions — trimebutine 3-thiocarbamoylbenzenesulfonate; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GIC-1001 oral tablets (Experimental): GIC-1001; 125 mg oral tablets; Single ascending doses (SAD) from 125 mg to 1000 mg; multiple ascending dose (MAD) from 125 mg to 500 mg TID over 7 successive days
  Interventions: Drug: GIC-1001; 125 mg oral tablets
- GIC-1001 matching placebo (Placebo Comparator): Matching placebo, single or multiple dosing
  Interventions: Drug: GIC-1001 matching placebo

INTERVENTIONS:
Drug: GIC-1001; 125 mg oral tablets — Single ascending doses (SAD) from 125 mg to 1000 mg;
  Multiple ascending doses from 125 mg to 500 mg, TID over 7 successive days
  Other Names: hydrogen sulfide releasing opioid agonist
  Arms: GIC-1001 oral tablets
Drug: GIC-1001 matching placebo — Single ascending doses (SAD) [equivalent to active arm, 125 mg to 1000 mg]
  Multiple ascending doses, TID over 7 successive days [equivalent to the active arm, 125 mg to 500 mg]
  Other Names: Same tablet-based excipients, without GIC-1001 (active)
  Arms: GIC-1001 matching placebo

SUMMARY:
The objectives of this single center, randomized, double-blinded, placebo-controlled Phase I clinical study are to evaluate the safety and tolerability of five (5) single and four (4) multiple increasing oral doses of GIC-1001 compared to placebo, and to evaluate the pharmacokinetics of GIC-1001 following single and multiple-dose administration in 80 healthy, 18-50 years old male and female subjects. Moreover, the effect of food on the pharmacokinetics of GIC-1001 in healthy subjects will be assessed. This study is designed with an integrated, adaptive approach which allows the evaluation of single and multiples doses of GIC-1001 in a progressive, overlapped fashion.

DETAILED DESCRIPTION:
Each cohort of enrolled healthy volunteers will include a total of eight (8) subjects: Six (6) subjects randomized to the active GIC-1001 and two (2) subjects randomized to a matching placebo.

Part 1: Single Doses Cohort A: Single dose of 125 mg of GIC-1001 or placebo; Cohort B: Single dose of 250 mg of GIC-1001 or placebo; Cohort C: Single dose of 375 mg of GIC-1001 or placebo; Cohort D: Single dose of 500 mg of GIC-1001 or placebo; and Cohort E: Single dose of 1000 mg of GIC-1001 or placebo. Up to 21 blood samples will be obtained over a 36 hour period.

Part 2: Multiple Doses, three times a day (TID) during 7 consecutive days; Cohort F: Multiple doses of 125 mg of GIC-1001 or placebo; Cohort G: Multiple doses of 250 mg of GIC-1001 or placebo; Cohort H: Multiple doses of 375 mg of GIC-1001 or placebo; and Cohort I: Multiple doses of 500 mg of GIC-1001 or placebo. Up to 18 blood samples will be obtained over a 7 day period.

Part 3: one single dose of GIC-1001 to be selected for the Food Effect cross-over evaluation. A total of 16 blood samples will be obtained over a 36 hour period.

Physical exams, 24 hour cardiac monitoring, and a complete battery of biochemical and hematological lab tests will be done to assess the safety and tolerability of GIC-1001 in all dosing cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteer
2. A female volunteer must meet one of the following criteria:

   1. Participant is of childbearing potential and agrees to use one of the accepted contraceptive regimens from the screening visit until 2 months after the last drug administration.

      or
   2. Participant is of non-childbearing potential, defined as a female who had had a hysterectomy or tubal ligation, is clinically considered infertile or is in a menopausal state (at least 1 year without menses)
3. A male volunteer with sexual partners who are pregnant, possibly pregnant, or who could become pregnant must meet the following criterion: Participant agrees to use one of the accepted contraceptive regimens from first drug administration until 3 months after the last drug administration.
4. Volunteer aged of at least 18 years but not older than 50 years
5. Volunteer with a body mass index (BMI) greater than or equal to 18.50 and below 30 kg/m2
6. Non- or ex-smokers. An ex-smoker is defined as someone who completely stopped smoking for at least 6 months before day 1 of this study
7. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance
8. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, biochemistry, ECG and urinalysis)

Exclusion Criteria:

1. History of significant hypersensitivity to trimebutine, to sulfur containing drugs (e.g. Captopril) or any related products (including excipients of the formulation) as well as severe hypersensitivity reactions (like angioedema) to any drugs
2. Presence of significant gastrointestinal, liver/kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
3. History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability
4. Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
5. Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
6. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 200 msec, QRS <60 msec, QRS >110 msec and QTc > 440 msec) on the screening ECG or other clinically significant ECG abnormalities
7. Known presence of rare hereditary problems of galactose and /or lactose intolerance
8. Use of cysteine, methionine, and other sulfur containing amino acid supplements in the previous 7 days before day 1 of this study
9. Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
10. Any clinically significant illness in the previous 28 days before day 1 of this study
11. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before day 1 of this study
12. Any history of tuberculosis and/or prophylaxis for tuberculosis
13. Positive urine screening of ethanol and/or drugs of abuse
14. Positive results to HIV, HBsAg or anti-HCV tests
15. Females who are pregnant according to a positive serum pregnancy test
16. Volunteers who took an Investigational Product (in another clinical trial) or donated 50 mL or more of blood in the previous 28 days before day 1 of this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in physical status | 8 hours post- drug administration
  Safety and Tolerability Monitoring: changes from baseline in blood pressure, pulse rate, oxygen saturation of blood, and body temperature will be measured at 8 hours post drug administration.

SECONDARY OUTCOMES:
Pharmacokinetics | Up to 36 hours for single ascending doses; every day and up to 8 hour post last dose for multiple ascending doses
  Blood samples will be obtained over a 36 hour period in the single dose portion of the study and over 7 days, every morning prior to GIC-1001, as well as 8 hours post-last dose in the multiple dosing phase. Main absorption and disposition parameters using a non-compartmental approach will be measured.
  For GIC-1001 and its metabolites, the pharmacokinetic parameters of interest for the single dose regimens will be Cmax, AUC0-8, AUCT, AUC∞, Tmax, AUCT/∞, Kel, T½el, Cl/F and Vd/F. The parameters Cmax, AUC0-8, AUCT and AUC∞ will be dose-normalized, and their natural logarithm will be calculated. The pharmacokinetic parameters of interest for the multiple dose regimens will be Cmax, Tmax, AUCτ, Cmin, Cpds, Fluctuation and Swing. The parameters Cmax, AUCτ and Cmin will be dose-normalized, and the natural logarithm of Cmax, AUCτ, Cmin and Cpds of will be calculated. For hydrogen sulfide and thiosulfate, the pharmacokinetic parameters of interest will be Cmax, Tmax and AUC0-4.
Change in ECG recording | 3 hours post drug administration
  Safety and Tolerability Monitoring: In all cohorts, change from baseline of 12-lead ECG will be measured at 3 hours post-drug administration.
Cardiac monitoring | 23 hours post drug administration
  Safety and Tolerability Monitoring: During Single Ascending Dosing only, continuous cardiac monitoring will be performed from approximately 1 hour prior to drug administration until at least 23 hours post-dose.
  In cases where the alarm activation of the monitoring system takes place for notification of concerns and/or rhythm changes, a rhythm strip will be printed and filed as source data. These occurrences will be followed up through further medical investigation, and/or filing of AEs.
  Any interruption of the patient monitoring due to clinical activities or else will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma Inc., Montreal, Quebec, Canada

REFERENCES:
- [Derived] Paquette JM, Rufiange M, Iovu Niculita M, Massicotte J, Lefebvre M, Colin P, Telmat A, Ranger M. Safety, tolerability and pharmacokinetics of trimebutine 3-thiocarbamoylbenzenesulfonate (GIC-1001) in a randomized phase I integrated design study: single and multiple ascending doses and effect of food in healthy volunteers. Clin Ther. 2014 Nov 1;36(11):1650-64. doi: 10.1016/j.clinthera.2014.08.005. Epub 2014 Sep 15. PMID 25224876